CLINICAL TRIAL: NCT00004414
Title: Sincalide (Cholecystokinin Octapeptide) Versus Placebo in Neonates at High Risk for Developing Parenteral Nutrition Associated Cholestasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13306; UMMS-FDR001449
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-05

CONDITIONS: Cholestasis
Keywords: cholestasis; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Cholestasis; Gastrointestinal Diseases; Rare Diseases | interventions — Sincalide

INTERVENTIONS:
Drug: sincalide

SUMMARY:
OBJECTIVES: I. Compare conjugated bilirubin levels and serum bile acid levels in severely premature newborns on long term parenteral nutrition and given either sincalide or placebo.

II. Compare morbidity and mortality rates in this patient population. III. Evaluate ultrasonographic images of the hepatobiliary tree during and 1 to 2 years after the administration of sincalide or placebo to assess the development of biliary sludge and biliary stone formation.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, placebo controlled, double blind, multicenter study. Patients are stratified according to prematurity or surgical group.

Patients are randomized to receive either placebo or sincalide IV over 10 to 15 minutes every 12 hours until a total of 8 weeks of therapy is administered or greater than 50% of their nutrition is enteral.

Patients are followed for a maximum of 2 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Severely premature neonates (less than 1000 g at birth and estimated gestational age of no greater than 28 weeks) that require greater than 50% of caloric requirements by parenteral means within 7 days of birth OR Neonates with one or more of the following surgical conditions: Necrotizing enterocolitis Gastroschisis Severe jejunal-ileal atresia within 7 days of diagnosis --Prior/Concurrent Therapy-- Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics No other cardiovascular (thoracotomy) or major gastrointestinal surgery (laparotomy) during the newborn period Other: No prior or concurrent ursodeoxycholic acid No concurrent use of extracorporeal life support --Patient Characteristics-- Performance status: Not specified Hematopoietic: Not specified Hepatic: Conjugated bilirubin no greater than 1.0 mg/dL No primary or secondary liver disease No hepatic insufficiency as documented by either a biopsy with cirrhosis or elevated prothrombin time without evidence of systemic coagulopathy and no administration of an anticoagulant Renal: No renal failure as indicated by a progressive increase in creatinine levels Other: No hemodynamic instability No documented communicable infection (including infectious hepatitis or HIV) No metabolic pathway defect that is associated with liver dysfunction in the neonatal period including hereditary fructose intolerance, galactosemia due to transferase deficiency, and neonatal tyrosinemia

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252
Dates: Start 1997-09; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hillel Teitelbaum, Study Chair — University of Michigan
Locations (6):
- United States (6):
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of Michigan Medical School, Ann Arbor, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor University Medical Center, Dallas, Texas